CLINICAL TRIAL: NCT05647109
Title: Department of Obstetrics & Gynecology ，Peking University People's Hospital
Brief Title: Patient-derived Tumor-like Cell Clusters Predict Progesterone Sensitivity in Patients With Early Endometrial Cancer
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University (Other); Beihang University (Other)
Responsible Party: Principal Investigator, Wang Jianliu, Professor, Doctoral supervisor, Chief physician, Vice President, Peking University People's Hospital
Other Study IDs: 2022PHB409
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Endometrial Carcinoma Stage I; Atypical Endometrial Hyperplasia
Keywords: Progesterone; Patient-derived tumor-like cell clusters; Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — fresh residual tissue available through biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Set of training: A total of 148 patients with endometrial cancer and atypical endometrial hyperplasia were included in the training set of the prediction model. They were divided into progesterone sensitive group and progesterone insensitive group.
  Interventions: Other: No intervention
- Set of verification: A verification set of the prediction model was established, consisting of 96 patients with endometrial cancer and atypical endometrial hyperplasia.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
To construct a prediction model of progesterone sensitivity in patients with endometrial cancer treated with fertility preservation

DETAILED DESCRIPTION:
After diagnosed of early endometrial carcinoma (EEC) or atypical endometrial hyperplasia (AEH) by hysteroscopy, patients meet the study criteria will be enrolled.

Patients will receive MPA (Medroxyprogesterone acetate) 250-500mg or MA (megestrol acetate) 160-320mg by mouth daily. Then hysteroscopy will be used to evaluate the endometrial condition every 3 months, and intra-operative findings will be recorded. Hysteroscopy will continue until pathology confirms complete response. Complete response (CR) is defined as the reversion of endometrial atypical hyperplasia to proliferative or secretory endometrium; partial response (PR) is defined as regression to hyperplasia with or without atypic; stable disease (SD) is defined as the persistence of the disease; and progressive disease (PD) is defined as the appearance of higher pathological progression, or myometrial invasion, or extra-uterine metastasis. Continuous therapies will be needed in PR or SD. Patients with PD will be recommended for hysterectomy.

During each hysteroscopy, the intraoperative residual tissues were sent to the laboratory of College of Future Science and Technology of Peking University for culture as Patient-derived tumor-like cell clusters (PTC), and the content of lipids (lipid droplet size and cholesterol content) was measured by stimulated Raman scattering imaging and recorded. After collecting the data of 148 cases, the prediction model was constructed. Then the model is validated in the validation set composed of 96 new cases. In order to determine the accuracy and sensitivity of the model.

If a patient has achieved a pathological complete response and a high lipid content is detected in the tissue by stimulated Raman scattering imaging, we will follow up for subsequent recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed pathological diagnosis based upon hysteroscopy: atypical endometrial hyperplasia or histologically prove well-differentiated EEC G1 without myometrial invasion
* No signs of suspicious extrauterine involvement on enhanced magnetic resonance imaging (MRI) or enhanced computed tomography (CT) or ultrasound
* Have a desire for remaining reproductive function or uterus
* Good compliance with adjunctive treatment and follow-up

Exclusion Criteria:

* Acute liver disease or liver tumor (benign or malignant) or renal dysfunction
* Pregnancy or potential pregnancy
* Confirmed diagnosis of any cancer in reproductive system
* Acute severe disease such as stroke or heart infarction or a history of thrombosis disease
* Hypersensitivity or contradiction for using MPA or MA
* With other factors of reproductive dysfunction;
* Strong request for uterine removal or other conservative treatment

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study focused on young, pre-menopausal patients with atypical endometrial hyperplasia or endometrioid adenocarcinoma diagnosed by hysteroscopic biopsy, who had a strong desire to preserve reproductive function.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
sensitivity | 7 months
  The sensitivity of the prediction model
accuracy | 7 months
  The accuracy of the prediction model

SECONDARY OUTCOMES:
false-negative rate | 7 months
  The false-negative rate of the prediction model
false-positive rate | 7 months
  The false-positive rate of the prediction model

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No